CLINICAL TRIAL: NCT01775904
Title: A Comparison Study of Capsule and Orally Disintegrating Tablet and to Determine the Effect of Food and Water on the Pharmacokinetics of LY2886721 in Healthy Subjects
Brief Title: A Study of Two Dosage Forms of LY2886721 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14249; I4O-MC-BACG (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — N-(3-(2-amino-4a,5,7,7a-tetrahydro-4H-furo(3,4-d)(1,3)thiazin-7a-yl)-4-fluorophenyl)-5-fluoropicolinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2886721 Capsule (water, fasting) (Experimental): Reference formulation. A single oral dose of 70 milligrams (mg) LY2886721 in a capsule given with water and without a meal in one of four periods.
  Interventions: Drug: LY2886721 in a Capsule
- LY2886721 ODT (no water, fasting) (Experimental): A single oral dose of 70 mg LY2886721 in an orally disintegrating tablet (ODT) given without water and without a meal in one of four periods.
  Interventions: Drug: LY2886721 in an orally disintegrating tablet (ODT)
- LY2886721 ODT (water, fed) (Experimental): A single oral dose of a 70 mg LY2886721 in an orally disintegrating tablet (ODT) given with water and after a high-fat breakfast in one of four periods.
  Interventions: Drug: LY2886721 in an orally disintegrating tablet (ODT)
- LY2886721 ODT (water, fasting) (Experimental): A single oral dose of 70 mg LY2886721 in an orally disintegrating tablet (ODT) given with water and without a meal in one of four periods.
  Interventions: Drug: LY2886721 in an orally disintegrating tablet (ODT)

INTERVENTIONS:
Drug: LY2886721 in a Capsule — Administered orally.
  Arms: LY2886721 Capsule (water, fasting)
Drug: LY2886721 in an orally disintegrating tablet (ODT) — Administered orally.
  Arms: LY2886721 ODT (no water, fasting); LY2886721 ODT (water, fasting); LY2886721 ODT (water, fed)

SUMMARY:
The purpose of this study is to evaluate two different formulations of LY2886721. In addition, this study will determine how much of study drug (LY2886721) gets into the blood steam and how long the body takes to get rid of it after taking each formulation with or without a meal. Information about any side effects that may occur will also be collected. Each participant may be involved in the study for approximately 7 weeks.

This study requires 4 periods. In each period, participants will receive LY2886721 as a tablet or capsule, with or without food and water. There is a 7 day washout between each period.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of 18.5 to 32.0 kilograms per square meter (kg/m^2), inclusive, at screening
* At least 4 participants who are greater than 55 years of age
* Male participants: Agree to use a reliable method of birth control and not donate sperm during the study and for 3 months following the last dose of the investigational product
* Female participants: Women not of child-bearing potential due to surgical sterilization (at least 6 weeks after surgical bilateral oophorectomy, hysterectomy, or both) confirmed by medical history, or postmenopausal females, as determined by medical history and physical examination (spontaneous amenorrhea for 6 to 12 months and a follicle stimulating hormone [FSH] level greater than 40 milli-international units per milliliter [mIU/mL])
* Have venous access sufficient to allow for blood sampling as per the protocol

Exclusion Criteria:

* Are currently enrolled in, have completed, or discontinued within the last 30 days from a clinical trial involving an investigational product; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated, within the last 30 days, in a clinical trial involving an investigational product
* Have known allergies to LY2886721, related compounds, or any components of the formulation
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* Have a significantly abnormal blood pressure as determined by the investigator
* Have a history or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis B or C and/or positive hepatitis B or C antibody
* Have a history of, or current, significant ophthalmologic disease
* Show evidence of significant active neuropsychiatric disease or history of suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Study Population: All participants who entered the study and received at least 1 dose of study drug.
Period: LY2886721 ODT (no Water, Fasting)
Arm/Group | Total Study Population
Started | 26
Received at Least One Dose of Drug | 26
Completed | 26
Not Completed | 0
Period: First Washout (7 Days)
Arm/Group | Total Study Population
Started | 26
Completed | 26
Not Completed | 0
Period: LY2886721 Capsule (Water, Fasting)
Arm/Group | Total Study Population
Started | 26
Received at Least One Dose of Drug | 26
Completed | 25
Not Completed | 1
Not completed — Adverse Event | 1
Period: Second Washout (7 Days)
Arm/Group | Total Study Population
Started | 25
Completed | 25
Not Completed | 0
Period: LY2886721 ODT (Water, Fed)
Arm/Group | Total Study Population
Started | 25
Received at Least One Dose of Drug | 25
Completed | 25
Not Completed | 0
Period: Third Washout (7 Days)
Arm/Group | Total Study Population
Started | 25
Completed | 25
Not Completed | 0
Period: LY2886721 ODT (Water, Fasting)
Arm/Group | Total Study Population
Started | 25
Received at Least One Dose of Drug | 24 (One participant was not dosed in this period due to an adverse event (AE).)
Completed | 24
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- Overall: All participants who entered the study and received at least 1 dose of study drug.
Arm/Group | Overall
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY2886721
Time Frame: Baseline through 96 hours post-dose
Population: Participants who received at least one dose of study drug with evaluable LY2886721 Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms / milliliter (ng/mL)
Groups:
- LY2886721 Capsule (Water, Fasting): A single oral dose of 70 milligrams (mg) LY2886721 in a capsule given with water and without a meal in one of four periods. Participants received a dose on the morning of Day 1 in each period. Participants were discharged on Day 5 of each period after study assessment. There was a washout period of at least 7 days between dosing in consecutive periods.
- LY2886721 ODT (no Water, Fasting): A single oral dose of 70 mg LY2886721 in an orally disintegrating tablet (ODT) given without water and without a meal in one of four periods. Participants received a dose on the morning of Day 1 in each period. Participants were discharged on Day 5 of each period after study assessment. There was a washout period of at least 7 days between dosing in consecutive periods.
- LY2886721 ODT (Water, Fed): A single oral dose of 70 mg LY2886721 in an ODT given with water and after a high-fat breakfast in one of four periods. Participants received a dose on the morning of Day 1 in each period. Participants were discharged on Day 5 of each period after study assessment. There was a washout period of at least 7 days between dosing in consecutive periods.
- LY2886721 ODT (Water, Fasting): A single oral dose of 70 mg LY2886721 in an ODT given with water and without a meal in one of four periods. Participants received a dose on the morning of Day 1 in each period. Participants were discharged on Day 5 of each period after study assessment. There was a washout period of at least 7 days between dosing in consecutive periods.
Arm/Group | LY2886721 Capsule (Water, Fasting) | LY2886721 ODT (no Water, Fasting) | LY2886721 ODT (Water, Fed) | LY2886721 ODT (Water, Fasting)
Number analyzed (Participants) | 26 | 26 | 25 | 24
nanograms / milliliter (ng/mL) | 183 (46) | 195 (29) | 181 (18) | 173 (37)

2. Primary Outcome: Pharmacokinetics (PK): Time of Maximum Observed Drug Concentration (Tmax) of LY2886721
Time Frame: Baseline through 96 hours post-dose
Population: Participants who received at least one dose of study drug with evaluable LY2886721 tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | LY2886721 Capsule (Water, Fasting) | LY2886721 ODT (no Water, Fasting) | LY2886721 ODT (Water, Fed) | LY2886721 ODT (Water, Fasting)
Number analyzed (Participants) | 26 | 26 | 25 | 24
hours | 3.00 [1.00 to 24.00] | 2.00 [1.00 to 4.00] | 4.00 [3.00 to 6.00] | 2.00 [1.00 to 12.00]

3. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Time Tlast (AUC[0-tlast]) of LY2886721
Time Frame: Baseline through 96 hours post-dose
Population: Participants who received at least one dose of study drug with evaluable LY2886721 AUC (0-tlast) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms * hour / milliliter
Arm/Group | LY2886721 Capsule (Water, Fasting) | LY2886721 ODT (no Water, Fasting) | LY2886721 ODT (Water, Fed) | LY2886721 ODT (Water, Fasting)
Number analyzed (Participants) | 26 | 26 | 25 | 24
nanograms * hour / milliliter | 2300 (24) | 2380 (19) | 2480 (19) | 2270 (18)

4. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞] of LY2886721
Time Frame: Baseline through 96 hours post-dose
Population: Participants who received at least one dose of study drug with evaluable LY2886721 AUC (0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms * hour / milliliter
Arm/Group | LY2886721 Capsule (Water, Fasting) | LY2886721 ODT (no Water, Fasting) | LY2886721 ODT (Water, Fed) | LY2886721 ODT (Water, Fasting)
Number analyzed (Participants) | 26 | 26 | 25 | 24
nanograms * hour / milliliter | 2320 (24) | 2390 (19) | 2490 (19) | 2290 (18)

ADVERSE EVENTS:
Arm/Group | LY2886721 Capsule (Water, Fasting) | LY2886721 ODT (no Water, Fasting) | LY2886721 ODT (Water, Fed) | LY2886721 ODT (Water, Fasting)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 9/26 | 8/26 | 6/25 | 7/24
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2886721 Capsule (Water, Fasting) (N=26) | LY2886721 ODT (no Water, Fasting) (N=26) | LY2886721 ODT (Water, Fed) (N=25) | LY2886721 ODT (Water, Fasting) (N=24)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Application site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 4 (4) | 2 (2) | 1 (1) | 2 (2)
Application site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days